CLINICAL TRIAL: NCT00530062
Title: Comparison of Single-Dose Efficacy of Albuterol-HFA-BAI and Albuterol-HFA-MDI in Asthmatics With Poor Inhaler Coordinating Ability
Brief Title: Comparison of Single-Dose Efficacy of an Albuterol Breath-Actuated Inhaler (Albuterol-HFA-BAI) Versus an Albuterol Metered-Dose Inhaler (Albuterol-HFA-MDI) in Participants With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IXR-404-04-167
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: Asthma and Poor Coordinators of Asthma Inhalers
MeSH Terms: conditions — Asthma | interventions — Albuterol; Procaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albuterol-HFA-BAI (Experimental): Participants will receive single actuation of albuterol 90 micrograms (mcg), administered using BAI in treatment period 1 or 2.
  Interventions: Drug: Albuterol-HFA-BAI
- Albuterol-HFA-MDI (Active Comparator): Participants will receive single actuation of albuterol 90 mcg, administered using MDI in treatment period 1 or 2.
  Interventions: Drug: Albuterol-HFA-MDI

INTERVENTIONS:
Drug: Albuterol-HFA-MDI — Inhalation Aerosols, 90 mcg, 1 dose per treatment period
  Other Names: Albuterol; ProAir
  Arms: Albuterol-HFA-MDI
Drug: Albuterol-HFA-BAI — Inhalation Aerosol (Breath-Actuated), 90 mcg, 1 dose per treatment period.
  Other Names: Albuterol
  Arms: Albuterol-HFA-BAI

SUMMARY:
This is a research study designed to compare the single-dose efficacy of albuterol-hydrofluoroalkane-breath-actuated inhaler (HFA-BAI) and albuterol-HFA-metered-dose inhaler (MDI) in asthmatics with poor inhaler coordinating abilities.

ELIGIBILITY:
Inclusion Criteria:

* Asthma of a minimum of 6 months duration
* Participants who demonstrate poor inhalation/actuation coordination when evaluated at screening utilizing the Aerosol Inhalation Monitor (AIM, Vitalograph) prior to any training and following training in 3 consecutive attempts
* Reversible bronchoconstriction of >12% increase in FEV1 with a cumulative dose of 450 mcg of albuterol
* The reversibility (FEV1) of ≤70% following administration of the initial 90 mcg of albuterol
* Ability to perform spirometry reproducibly
* Ability to self-perform peak expiratory flow (PEF) determinations and report scores on diaries
* Can tolerate withdrawal of applicable medications for qualification at screening
* Otherwise healthy individuals
* Non-smokers for at least 2 years prior to the screening visit

Exclusion Criteria:

* Allergy or sensitivity to albuterol
* Exposure to investigational drugs within 30 days prior to the screening visit
* Continuous treatment with beta-blockers, monoamine oxidase (MAO) inhibitors, tricyclic antidepressants, and/or systemic corticosteroids
* Treated with oral or injectable corticosteroids within the 6 weeks prior to the screening visit
* The prescribed dose regimen of any required antileukotrienes, inhaled corticosteroids and/or inhaled cromolyn and/or nedocromil had not been stable for at least 4 weeks prior to the screening visit
* Inability to tolerate or unwillingness to comply with required washout periods for all applicable medications
* Hospitalization for acute exacerbation of asthma more than twice in past year
* Treatment in an emergency room or hospitalization for asthmatic symptoms within 3 months prior to the screening visit
* An upper respiratory tract infection and/or sinusitis associated with exacerbation of asthma that is unresolved 3 weeks prior to the screening visit
* History and/or presence of any clinically significant non-asthmatic acute or chronic disease
* Known or suspected substance abuse
* Previous enrollment in an IVAX Research-sponsored Albuterol-HFA asthma study Note: Other inclusion and exclusion criteria may apply.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-07-25 (Actual); Primary Completion 2008-10-24 (Actual); Study Completion 2008-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (5):
- United States (5):
  - Clinical Study Site, Huntington Beach, California
  - Teva Clinical Study Site, Lakewood, Colorado
  - Clinical Study Site, Minneapolis, Minnesota
  - Clinical Study Site, Oklahoma City, Oklahoma
  - Clinical Study Site, Lake Oswego, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized to receive the following 2 treatments on separate occasions 2-7 days apart: Albuterol-hydrofluoroalkane-breath-actuated inhaler (HFA-BAI) and Albuterol-HFA-metered-dose inhaler (MDI).
Groups:
- Overall Population: Participants received single actuation of albuterol 90 micrograms (mcg), administered using BAI in treatment period 1, then single actuation of albuterol 90 mcg, administered using MDI in treatment period 2. There was a washout period of 2-7 days between treatments.
Period: Overall Study
Arm/Group | Overall Population
Started | 49
Received at Least 1 Dose of Study Drug | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of the assigned study medication.
Groups:
- Overall Population: Participants received single actuation of albuterol 90 mcg, administered using BAI in treatment period 1, then single actuation of albuterol 90 mcg, administered using MDI in treatment period 2. There was a washout period of 2-7 days between treatments.
Arm/Group | Overall Population
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African heritage | 2
  Race: White | 47

OUTCOME MEASURES:

1. Primary Outcome: Area-Under-the-Effect Curve of Percent Change in Test-Day Baseline Forced Expiratory Volume in 1 Second (FEV1) Versus Time (up to 2 Hours Postdose), %FEV1 AUEC0-2
Description: The %FEV1 AUEC0-2 was calculated using the linear trapezoidal rule. The baseline value consisted of the average of the two predose FEV1 measurements. The mean was obtained from the mixed-effect analysis of variance adjusted for effects from the study center, the treatment sequence, and study period.
Time Frame: Baseline, Up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Mean (Standard Error); unit: percent change from baseline*hour
Groups:
- Albuterol-HFA-BAI: Participants received single actuation of albuterol 90 mcg, administered using BAI in treatment period 1
- Albuterol-HFA-MDI: Participants received single actuation of albuterol 90 mcg, administered using MDI in treatment period 2.
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
percent change from baseline*hour | 21.403 (2.263) | 20.457 (2.253)
Statistical Analysis 1: Comparison: Albuterol-HFA-BAI vs Albuterol-HFA-MDI; The analysis was performed using the mixed-effect analysis of variance with fixed effects of center, sequence, treatment group and period, and random effect of the participant within sequence; Test type: Other; p = 0.5595, ANCOVA — Threshold for significance at 0.05 level; Difference in adjusted mean = 0.946, 95% CI 2-sided [-2.293 to 4.185]

2. Secondary Outcome: Percent Change From Baseline in FEV1 Within 30 Minutes Postdose
Description: The mean was obtained from the mixed-effect analysis of variance adjusted for effects from the study center, the treatment sequence, and study period.
Time Frame: Baseline up to 30 minutes postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
percent change | 10.777 (1.185) | 10.114 (1.180)

3. Secondary Outcome: Percent Change From Baseline in FEV1 up to 2 Hours Postdose
Description: as for outcome 2
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
percent change | 14.319 (1.292) | 13.731 (1.286)

4. Secondary Outcome: Area-Under-the-Effect Curve of Change in Test-Day Baseline FEV1 Versus Time (up to 2 Hours Postdose), FEV1 AUEC0-2
Description: The %FEV1 AUEC0-2 was calculated using the linear trapezoidal rule. The test-day baseline consisted of the average of the two predose FEV1 measurements. The mean was obtained from the mixed-effect analysis of variance adjusted for effects from the study center, the treatment sequence, and study period.
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Mean (Standard Error); unit: liters*hours
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
liters*hours | 0.443 (0.044) | 0.407 (0.044)

5. Secondary Outcome: Percentage of Participants With a 12% Increase From Baseline in FEV1 Within 2 Hours Postdose
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
percentage of participants | 57.1 | 42.9

6. Secondary Outcome: Percentage of Participants With a 15% Increase From Baseline in FEV1 Within 2 Hours Postdose
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
percentage of participants | 32.7 | 30.6

7. Secondary Outcome: Time to a 12% Increase From Baseline in FEV1 Within 2 Hours Postdose
Description: The number of minutes required for the baseline FEV1 to increase by at least 12% within the 2-hour observation period. Median time and corresponding confidence intervals (CIs) were obtained via the Kaplan-Meier estimate.
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
minutes | 60.00 [45.00 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI was not estimable. | NA [46.00 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI was not estimable.

8. Secondary Outcome: Time to a 15% Increase From Baseline in FEV1 Within 2 Hours Postdose
Description: The number of minutes required for the baseline FEV1 to increase by at least 15% within the 2-hour observation period. Median time and corresponding CIs were obtained via the Kaplan-Meier estimate.
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
minutes | NA [123.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI was not estimable. | NA [NA to NA] — Not enough participants experienced a 15% increase in FEV1 and therefore the median could not be calculated.

9. Secondary Outcome: Time to Maximum Increase in FEV1
Description: Each calculation for FEV1 took several minutes in order to obtain the highest of 3 measurements. The total collection time exceeded the 120 mins post-dose time frame for some participants.
Time Frame: Baseline up to 2 hours postdose
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication.
Measure: Median (Full Range); unit: minutes
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
Number analyzed (Participants) | 49 | 49
minutes | 48.00 [15.00 to 123.0] | 45.00 [11.00 to 128.0]

ADVERSE EVENTS:
Time Frame: From the day of study drug administration up to 30 days
Description: Safety population included all randomized participants who took at least 1 dose of the assigned study medication.
Arm/Group | Albuterol-HFA-BAI | Albuterol-HFA-MDI
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.